CLINICAL TRIAL: NCT06729567
Title: Number of Dermatomes Blocked by Conventional Dose Single Shot Spinal Anaesthesia for Cesarean Section May Not be Related to Hyperbaric Bupivacaine Dose - a Retrospective Analysis.
Brief Title: Dose-to-block Level Relation in Single Shot Spinal Anesthesia for Cesarean Section.
Acronym: SpinDoBlock
Status: Active, not recruiting | Type: Observational
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Principal Investigator, Bartosz Horosz, MD, Principal Investigator, Centre of Postgraduate Medical Education
Other Study IDs: 97/2024
Record Dates: First submitted 2024-12-01; First posted 2024-12-11 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Spinal Anesthesia Evaluation; Cesarean Delivery
Keywords: spinal anesthesia; cesarean section; spinal block level
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients given spinal block with conventional dose of bupivacaine for cesarean delivery: Using electronic hospital database we will identify cases of cesarean section. Initially, all cases of cesarian delivery under spinal anesthesia will be identified. After that, manual review of the anesthetic charts will follow. Detailed data on anesthetic technique will be retrieved and cases where conventional dose of hyperbaric bupivacaine was used will be included in further analysis. Further review of the charts will provide demographic data of the parturients, data on vital signs during anesthesia and dynamic of sensory block level. Attention will be paid to assure that identification of the patient would not be possible with data used in this study. All identifiable data used in data retrieval process and analysis will be accessible only for investigators.
  Interventions: Other: Spinal block level analysis; Other: data collection

INTERVENTIONS:
Other: Spinal block level analysis — Relation of the dose of hyperbaric bupivacaine to resulting spinal block level is to be assessed. Conventional dose cases (more than 9mg and less than 13mg) will be included in analysis.
Other: data collection — Intervention is to acquire and analyse anonymous perioperative data. After identification of the eligible cases, statistical analysis will be performed.

SUMMARY:
The study is designed to support or deny relation between the dose of hyperbaric bupivacaine given intrathecally and extent of spinal block level. There is ongoing debate whether anesthetists should adjust the dose in the range of conventional doses in order to achieve appropriate coverage of anesthesia which would be suitable for cesarean section.

Two strategies are predominantly used: low dose strategy, which is focused on safety, and conventional dose approach, which is more effective in terms of success of anesthesia, with markedly higher rate of spinal block - related complications. It is hypothesized that there may be no relation between block level and the dose if conventional doses are used. For that purpose anesthetic charts of cesarean sections will be reviewed to gather information on the doses of anesthetic used and the level of spinal block they produced.

DETAILED DESCRIPTION:
Single - shot spinal block for cesarean delivery is a gold standard in obstetric anesthesia. Both level and density of the block may have direct impact on the quality of surgery, patient's comfort and the course of postoperative recovery. Ideal dose of local anaesthetic for single - shot spinal anesthesia is still to be decided, with ongoing debate on using either "low" or "conventional" doses as routine approach. Use of conventional doses of local anesthetic (doses nearing dose effective in 95 percent of patients,ED95) have proven to be superior to low dose regimens in terms of effectiveness and therefore this strategy is widely used, despite the higher risk of spinal block - related complications.

Amount of local anesthestic used is regarded to be a factor of significant influence on its intrathecal spread and the final level of block following single - shot spinal anesthesia. It was investigated in both general and obstetric populations, although most of the studies with results in favor of this relation were designed to assess the other factors, and the extend of sensory block was not set as their primary outcome.

It was previously reported that adjusting the conventional dose of hyperbaric bupivacaine to parturient's height does not change the risk of block failure and rate of complications when compared to fixed - dose regimen. Whether the change in bupivacaine dose within the range of conventional doses results in significant change in sensory block level is not clear.

This retrospective analysis was designed to assess the above relation

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery at term under spinal anesthesia
* American Society of Anesthesiologists (ASA) physical status <3
* BMI<40

Exclusion Criteria:

* Spinal anesthesia with less than 9mg of hyperbaric bupivacaine
* Local anesthetic other than hyperbaric bupivacaine used
* Failed spinal anesthesia
* Poor quality of the anesthetic record - data required for analysis not available

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Initial cohort for the study will be selected from the cases of cesarean section in years 2017 - 2022, who delivered in Orlowski Hospital, Department of Obstetrics and Gynaecology, Warsaw, Poland. Intention is to include at least 300 participants in the final analysis, to allow for regression analysis.
Sampling Method: Non-Probability Sample
Enrollment: 362 (Actual)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Dose - extent correlation coefficient | Highest level of sensory block noted from the time of spinal injection until the end of surgical procedure
  Pearson's and/or Spearman's correlation coefficient will be employed to asses relation between the dose and level of the sensory block. For the purpose of analysis the extent of the block will be expressed as a number of blocked dermatomes (S-5, L-5, T-12,C-8) for more reliable statistical analysis. Regression analysis will be performed if significant relation is found.

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Malec-Milewska, MD, Prof., Study Chair — Department of Anesthesia and Intensive Care, Orlowski Hospital, Warsaw
Locations (1):
- Department of Anesthesiology and Intensive Care, Centre of Postgraduate Medical Education, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ozkan Seyhan T, Orhan-Sungur M, Basaran B, Savran Karadeniz M, Demircan F, Xu Z, Sessler DI. The effect of intra-abdominal pressure on sensory block level of single-shot spinal anesthesia for cesarean section: an observational study. Int J Obstet Anesth. 2015 Feb;24(1):35-40. doi: 10.1016/j.ijoa.2014.08.004. Epub 2014 Aug 27. PMID 25499016
- [Background] Visavakul O, Leurcharusmee P, Pipanmekaporn T, Khorana J, Patumanond J, Phinyo P. Effective Dose Range of Intrathecal Isobaric Bupivacaine to Achieve T5-T10 Sensory Block Heights for Elderly and Overweight Patients: An Observational Study. Medicina (Kaunas). 2023 Mar 1;59(3):484. doi: 10.3390/medicina59030484. PMID 36984485
- [Background] Huang YY, Chang KY. Sensory block level prediction of spinal anaesthesia with 0.5% hyperbaric bupivacaine: a retrospective study. Sci Rep. 2021 Apr 27;11(1):9105. doi: 10.1038/s41598-021-88726-2. PMID 33907264